CLINICAL TRIAL: NCT00621803
Title: Prevention of Gastric Colonisation by Antibiotic Resistant Pseudomonas Aeruginosa Strains Using Oral Probiotic in ICU-Patients
Brief Title: Lcr35 / ICU / P. Aeruginosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting or enrolling participants has halted and will not resume
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Christophe De Champs, Chu Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0029; AFSSAPS 1220/CM/FE02
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Pseudomonas Infections
Keywords: Probiotic; Pseudomonas aeruginosa; Gastric colonization; Respiratory tract colonization; Ventilator aquired pneumoniae; determine the effect of oral administration of this probiotic on gastric and respiratory tract colonisation/infection by P. aeruginosa
MeSH Terms: conditions — Pseudomonas Infections

INTERVENTIONS:
Drug: Probiotic Lactobacillus casei rhamnosus (Lcr35)

SUMMARY:
Preventing carriage of potentially pathogenic micro-organisms from the aerodigestive tract is an infection control strategy used to reduce the occurrence of nosocomial infections - including ventilator-assisted pneumonia - in intensive care units. The use of antibiotics is controversial and can lead to adverse effect such as the selection of highly resistant pathogens. The purpose of this study was to investigate the effect of oral administration of a probiotic strain, Lactobacillus, on gastric and respiratory tract colonisation/infection by Pseudomonas aeruginosa strains, according to the concept that an indigenous flora has a protective effect against secondary colonisation.

DETAILED DESCRIPTION:
In this prospective double-blind randomised study, ICU patients receive twice a day either an oral dose of Lactobacillus casei rhamnosus, the available pharmaceutical form, or a placebo. Digestive tract carriage of Pseudomonas aeruginosa is monitored by cultures of gastric aspirates. The occurrence of respiratory tract colonisations / infections is monitored throughout the study. Evaluation criteria are the delay and the rates of gastric P. aeruginosa colonisation and respiratory tract infection or colonisation. Chi-square or two tailed Fisher exact test are used for comparing qualitative variables and Student's t-test or mann-Whitney test for quantitatives variables. The mean of non-acquisition expectancy (NAE), length of stay without P. aeruginosa acquisition, was calculated and P. aeruginosa non-colonized patient rates were estimated and the two groups compared with regard to survival curves from grouped data using the Kaplan Meier method and the Logrank test. Variables with a P. value ≤0.15 in the univariate analysis were included in a logistic regression and a Cox regression model for multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* length of stay longer than 48h
* with a nasogastric feeding tube

Exclusion Criteria:

* - less than 18 years old
* length of stay < 48h
* immunosuppression
* absolute neutrophile count < 500/mm3
* gastro-intestinal bleeding
* contraindicated enteral feeding
* positive P. aeruginosa gastric aspirates or respiratory tract specimens during the first four days after hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2003-03; Primary Completion 2004-10 (Estimated); Study Completion 2005-10 (Estimated)

PRIMARY OUTCOMES:
Delay in P.aeruginosa colonisation

SECONDARY OUTCOMES:
Delay of respiratory tract infection or colonisation due to P.aeruginosa. Persistance of L.casei rhamnosus in to the stomach

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Champs, MD PhD, Principal Investigator — University Hospital, Clermont-Ferrand